CLINICAL TRIAL: NCT01713426
Title: Qutenza Versus Pregabalin in Subjects With Peripheral Neuropathic Pain: an Open-label, Randomized, Multicenter, Non-inferiority Efficacy and Tolerability Study
Brief Title: A Study to Compare QUTENZA With Pregabalin for the Treatment of Peripheral Neuropathic Pain (PNP) After 8 Weeks of Treatment
Acronym: ELEVATE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Europe Ltd. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QTZ-EC-0004; 2011-005872-41 (EudraCT Number)
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2018-04-23 (Actual); Status verified 2018-04

CONDITIONS: Non-diabetic Painful Peripheral Polyneuropathy; Postherpetic Neuralgia (PHN); Peripheral Nerve Injury (PNI)
Keywords: Post herpetic neuralgia; Qutenza; NGX-4010; Peripheral Neuropathic Pain; Pregabalin
MeSH Terms: conditions — Neuralgia, Postherpetic; Peripheral Nerve Injuries | interventions — Capsaicin; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Qutenza (Experimental): Cutaneous patch
  Interventions: Drug: Qutenza
- Pregabalin (Active Comparator): Oral capsule
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Qutenza — Cutaneous patch
  Other Names: Capsaicin
  Arms: Qutenza
Drug: Pregabalin — Oral capsule
  Arms: Pregabalin

SUMMARY:
This study is comparing the efficacy and tolerability of Qutenza with that of pregabalin in patients suffering from peripheral neuropathic pain. Treatment allocation will be to one of these treatments and the duration of the study will be about 10 weeks (assuming that from screening to treatment allocation takes 2 weeks). Participants will be asked to complete questionnaires about various aspects relating to their condition throughout the study.

This study will include subjects suffering from Postherpetic Neuralgia, Peripheral Nerve Injury or Non Diabetic peripheral polyneuropathy.

ELIGIBILITY:
Inclusion Criteria:

* 1. Documented diagnosis of probable or definite PNP
* 2. Localized and well-defined area of PNP, suitable for treatment with QUTENZA
* 3. Documented diagnosis at the Baseline Visit of either:

  * Postherpetic neuralgia (PHN) with pain persisting at least 6 months since shingles vesicle crusting
  * Peripheral nerve injury (PNI) including post-surgical or post-traumatic neuropathic pain, persisting for a minimum of 3 months
  * Non-diabetic painful peripheral polyneuropathy with pain which has persisted for a minimum of 3 months, including (i) small-fiber neuropathy, as confirmed by quantitative sensory testing (QST), laser evoked potentials (LEP) or skin biopsy, (ii) chemotherapy induced neuropathy in subjects with stable neoplastic disease, (iii) other, adequately characterized painful peripheral polyneuropathy, based on clinical history and examination
* 4. Average pain score ≥4 during Screening Period, over a minimum of at least 4 consecutive days (using the "average pain for the past 24 hours" Numeric Pain Rating Scale (NPRS) score
* 5. Intact, non-irritated, dry skin over the painful area(s) to be treated
* 6. Is either:

  * Naïve to treatment with pregabalin and gabapentin, OR
  * In the opinion of the investigator, has not received an adequate trial of treatment with pregabalin or gabapentin
* 7. Subject is willing to receive pregabalin or QUTENZA as part of the trial
* 8. Females of child bearing potential must be willing to use highly effective methods of birth control during the study and for 30 days following study termination

Exclusion Criteria:

* 1. Significant ongoing or recurrent pain of etiology other than PHN, PNI or non-diabetic painful peripheral polyneuropathy, for example: compression-related neuropathies (e.g. spinal stenosis), radiculopathy, tumor-related pain, fibromyalgia or arthritis
* 2. Complex Regional Pain Syndrome (CRPS, Type I or II)
* 3. Neuropathic pain related to previously administered radiotherapy, diabetes mellitus or HIV-AN
* 4. Neuropathic pain areas located only on the face, above the hairline of the scalp, and/or in proximity to mucous membranes
* 5. Severe loss of heat sensation in the painful area, indicative of C-fiber denervation
* 6. Reported daily pain score of 10 on the NPRS for at least 4 days during the Screening Period
* 7. Past or current history of diabetes mellitus
* 8. Unstable or poorly controlled hypertension or a recent history of a cardiovascular event which, in the opinion of the investigator, would put the subject at risk of adverse cardiovascular reactions related to the patch application procedure
* 9. Creatinine clearance (CLcr) < 60mL/min according to the Cockcroft-Gault formula
* 10. Untreated ongoing generalized anxiety disorder according to DSM-IV or ICD-10 criteria
* 11. Severe ongoing depression according to DSM-IV or ICD-10 criteria
* 12. Evidence of cognitive impairment including dementia that may interfere with subject's ability to complete study evaluations and recall pain levels in the past 24 hours
* 13. Planned elective surgery during the trial
* 14. Changes to stable neuropathic pain background medication in the 4 weeks prior to the Baseline Visit
* 15. Any prior receipt of QUTENZA patches, including blinded patches administered as part of a clinical trial
* 16. Hypersensitivity to capsaicin (i.e., chilli peppers or Over-the-counter [OTC] capsaicin products), any QUTENZA excipients, local anesthetics, or adhesives
* 17. Treatment with pregabalin or gabapentin within 2 months prior to the Baseline Visit
* 18. Hypersensitivity to pregabalin or any of the excipients
* 19. Use of opioids exceeding a total daily dose of morphine of 200 mg/day, or equivalent; or any intravenous opioids or tapentadol, regardless of dose, within 7 days preceding the Baseline Visit
* 20. Use of any topical pain medication, such as non-steroidal anti-inflammatory drugs, menthol, methyl salicylate, local anesthetics (including patch containing lidocaine), steroids or capsaicin products on the painful areas to be treated within 7 days preceding the Baseline Visit
* 21. Chemotherapy within 3 months of the Baseline Visit, except maintenance hormone treatment
* 22. Use of any investigational agent within 30 days prior to Baseline Visit
* 23. Active substance abuse or history of chronic substance abuse within 1 year prior to screening; or any prior chronic substance abuse (including alcoholism) likely to re-occur during the study period as judged by the investigator
* 24. Female subjects of child-bearing potential with a positive serum or urine pregnancy test prior to treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Actual)
Dates: Start 2012-07-11 (Actual); Primary Completion 2013-09-26 (Actual); Study Completion 2013-09-26 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each arm who achieve at least 30% decrease in the "average pain for the past 24 hours" Numeric Pain Rating Scale (NPRS) score from baseline to week 8 | Baseline and week 8

SECONDARY OUTCOMES:
Proportion of subjects in each arm who achieve "optimal Therapeutic effect" | Baseline and week 8
  Optimal therapeutic effect is defined as:
  * No change in background chronic pain medication and no discontinuation of study drug due to lack of efficacy or tolerability prior to Week 8
  * At least a 30% reduction in the "average pain for the past 24 hours" NPRS score, from baseline to Week 8, and
  * No moderate or severe adverse drug reactions (ADRs) during the stable Treatment Period
Proportion of subjects who achieve at least a 30% decrease in the "average pain for the past 24 hours" | Baseline to Week 8
  NPRS score from baseline to the mean of all scores recorded between Week 1 (Day 8) and Week 8 (Day 57)
Proportion of subjects who achieve at least a 50% decrease in the "average pain for the past 24 hours" | Baseline to Week 8
  NPRS score from baseline to week 8, and from baseline to the mean of all scores recorded between Week 1 (Day 8) and Week 8 (Day 57)
Absolute and percent change in "average pain for the past 24 hours" | Baseline to Week 8
  NPRS score from baseline to Week 8, and from baseline to the mean of all scores recorded between Weeks 1 to 8
Time to onset of pain relief (in days) | Up to 8 weeks
  Assessed by at least a 30% reduction in "average pain for the past 24 hours" NPRS score
Overall subject status using Patient Global Impression of Change (PGIC) questionnaire | At Weeks 4 and 8
Change in the Medical Outcomes Study (MOS) 6-Item Cognitive Functioning Scale | Baseline to Week 8
MOS - Sleep Scale | Baseline to Weeks 4 and 8
Change in the EQ-5D-5L (Euroqol-5 dimensions-5 levels) total score | Baseline to Week 8
Treatment satisfaction | Baseline to Weeks 4 and 8
  As assessed by:
  * Proportion of subjects who discontinue study drug or withdraw from the study due to either a lack of efficacy or tolerability
  * Treatment Satisfaction Questionnaire for Medication (TSQM) questionnaire at Week 4 and Week 8
Treatment satisfaction - continuance of treatment | Week 8
  As assessed by willingness to continue treatment at Week 8
Time to reach optimal maintenance dose for pregabalin | Baseline to Week 8
Healthcare Resource use | Baseline to Week 8
  Number of contacts with health professionals
Tolerability (Assessed by the number, severity and duration of ADRs) | Baseline to Week 8
  Collected as self-rated health-related complaints by the subject and then medically confirmed and causality assigned by the investigator
Change in intensity and area of allodynia | Baseline to Week 8
Changes in sensory symptoms | Baseline to Week 8
  Assessed using Neuropathic Pain Symptom Inventory (NPSI) scores
Reduction in pain | Baseline to Week 8
  By the pattern of sensory symptoms as defined using NPSI scores at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe Ltd.
Locations (98):
- Armenia (4):
  - Site 101 Medical Union 2, Yerevan
  - Site 102 Medical Center Erebuni, Yerevan
  - Site 103 Scientific research Institute of physiotherapy, Yerevan
  - Site 104 Medical Center "Surb Nerses Mets", Yerevan
- Austria (5):
  - Site 114 Klinikum Klagenfurt Worthersee, Klagenfurt, Carynthia
  - Site 115 Medical University Innsbruck, Innsbruck, Tyrol
  - Site 116 Krankenhaus der Barmherzigen B, Graz
  - Site 111 AKH Universitatsklinik, Vienna
  - Site 112 Wilhelminenspital, Vienna
- Site 121 Vitebsk Regional Clinical Hospital # 1, Vitebsk, Belarus
- Belgium (7):
  - Site 131 UZ Brussels, Brussels
  - Site 138 Cliniques Universitaires Saint, Brussels
  - Site 134 Grand Hospital de Charleroi, Charleroi
  - Site 137 Univ. Ziekenhuis Antwerpen, Edegem
  - Site 132 Ziekenhuis Oost-Limburg, Genk
  - Site 136 UZ Pellenberg, Pellenberg
  - Site 133 Heilig Hart Ziekenhuis, Roeselare
- Bulgaria (6):
  - Site 142 UMHAT - Pleven, Pleven
  - Site 141 Centre for Mental Health, Rousse
  - Site 144 Tokuda Hospital Sofia, Sofia
  - Site 146 MHAT Alexandrovska Hospital, Sofia
  - Site 147 MHAT Sv. Ivan Rilski, Sofia
  - Site 145 Military Medical Academy, Sofia
- Czechia (2):
  - Site 151 Fakultni nemocnice Plzen, Pilsen
  - Site 153 Klinika anesteziologie, Prague
- Finland (3):
  - Site 163 ORTON Invalidisaatio, Helsinki
  - Site 161 Finnmedi OY, Tampere
  - Site 162 Vassa Central Hospital, Vaasa
- France (7):
  - Site 171 Hospital Ambroise Pare, Boulogne-Billancourt
  - Site 174 Hopital Neurologique Pierre W, Bron
  - Site 177 Hospital Roger Salengro CHRU, Lille
  - Site 175 CHU Caremeau, Nîmes
  - Site 172 Hospital Saint Antoine, Paris
  - Site 173 CHU Hopital Nord, Saint-Etienne
  - Site 176 CH Regional de Valence, Valence
- Germany (5):
  - Site 200 Prax S.Wolf u.B.Schütz Pal.med, Cottbus
  - Site 192 Universitätsklinikum Giessen, Giessen
  - Site 193 Universitätsklinikum Münster, Münster
  - Site 194 Schmerz Palliativznt Wiesbaden, Wiesbaden
  - Site 197 Universitätsklinikum Würzburg, Würzburg
- Greece (4):
  - Site 204 Athens Naval Hospital, Athens
  - Site 202 Hippokration General Hospital of Athens, Athens
  - Site 201 Aretaieio University Hospital, Athens
  - Site 203 Aretaieio/Maginio Hospital, Athens
- Site 213 Semmelweis Egyetem Molekuláris Neurológiai Klinikai és Kutatási Központ, Budapest, Hungary
- Italy (11):
  - Site 227 Azienda Ospedaliera Universita, Florence
  - Site 222 A.O.U Ospedali Riuniti, Foggia
  - Site 232 Ospedale Niguarda Ca' Granda, Milan
  - Site 225 Policlinico San Donato, Milan
  - Site 221 FONDAZIONE S.MAUGERI I.R.C.C.S, Pavia
  - Site 228 Azienda Ospedaliero di Perugia, Perugia
  - Site 229 Azienda Ospedaliero di Perugia, Perugia
  - Site 231 Ospedale S. Chiara, Pisa
  - Site 226 Presidio Ospedale G.Mazzini, Teramo
  - Site 230 Azienda Ospedaliera SantaMaria, Terni
  - Site 223 AOU San Giovanni Battista, Torino
- Poland (6):
  - Site 244 Niepubliczny Zakład Opieki Zdr, Gdansk
  - Site 245 Poradnia Leczenia Bólu, Uniwer, Gdansk
  - Site 243 NZOZ Poradnia Leczenia Bólu, Gdynia
  - Site 241 Tomasz Dąbrowski Śląskie Centr, Katowice
  - Site 246 NZOZ Poradnia Leczenia Bolu Pr, Tychy
  - Site 242 NZOZ Centrum Medyczne, Warsaw
- Portugal (3):
  - Site 254 Hospital Fernando Fonseca, Amadora
  - Site 252 Instituto Portuges de Oncologic, Lisbon
  - Site 253 CHS - Hosp. S. Bernardo, Setúbal
- Romania (6):
  - Site 261 Quantum Medical Center SRL, Bucharest
  - Site 264 Spitalul Clinic Colentina, Bucharest
  - Site 262 Spitalul Clinic Judetean de Ur, Constanța
  - Site 266 Spitalul Clinic de Urgenta "Pr, Iași
  - Site 265 Spit Clin Judetean de Urgenta, Târgu Mureş
  - Site 263 Spitalul Clinic Judetean de Ur, Timișoara
- Russia (7):
  - Site 271 First Moscow State Medical University named after I.M. Sechenov, Moscow
  - Site 272 City Clinical Hospital # 12, Moscow
  - Site 278 Semashko Regional Clinical Hospital, Nizhny Novgorod
  - Site 276 OOO Clinical Neurology Center, Novosibirsk
  - Site 273 Military Medical Academy, Saint Petersburg
  - Site 274 Saint-Petersburg State Medical University, Saint Petersburg
  - Site 277 Hospital №40 of Kurortniy, Saint Petersburg
- Slovakia (3):
  - Site 282 Neurological surgery, Bratislava
  - Site 281 AB-BA ambulancia, Bratislava
  - Site 283 SANERA, s.r.o., Prešov
- Site 292 University Medical Centre Mari, Maribor, Slovenia
- Spain (2):
  - Site 301 Hospital General Universitario de Alicante, Alicante
  - Site 303 Hospital Universitario Virgen, Granada
- Sweden (3):
  - Site 313 SU/Östra, Gothenburg
  - Site 311 Karolinska University Hospital, Stockholm
  - Site 312 Karolinska University Hospital, Stockholm
- Turkey (Türkiye) (5):
  - Site 321 Hacettepe University Medical Faculty Hospital, Ankara
  - Site 325 Pamukkale University Medical Faculty Hospital, Denizli
  - Site 326 Maramara University, Pendik Training and Research Hospital, Istanbul
  - Site 323 Ege University Medical Faculty Hospital, Izmir
  - Site 324 Dokuz Eylul University Medical Faculty Hospital, Izmir
- United Kingdom (6):
  - Site 332 Gartnavel General Hospital, Glasgow
  - Site 334 Seacroft Hospital, Leeds
  - Site 336 Leicester Royal Infirmary, Leicester
  - Site 331 The Walton Centre, Liverpool
  - Site 333 St Thomas' Hospital, London
  - Site 335 The Christies NHS Foundation, Manchester

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Viel E, Eerdekens M, Kandaswamy P. Treatment Impact on Patient-Reported Outcomes in Peripheral Neuropathic Pain: Comparing Single Intervention With Topical High-Concentration Capsaicin to Daily Oral Pregabalin. Pain Physician. 2021 Sep;24(6):453-463. PMID 34554688
- See also: Link to results on EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2011-005872-41/results
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/study.aspx?ID=83